CLINICAL TRIAL: NCT01930617
Title: Irrigation of Chronic Subdural Hematomas - is More Better? A Population Based Study Between Different Treatment Policies
Brief Title: Irrigation of Chronic Subdural Hematomas - is More Better?
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); University Hospital of North Norway (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/2050
Record Dates: First submitted 2013-08-22; First posted 2013-08-29 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Hematoma, Subdural, Chronic
Keywords: surgery; trephining; drainage; therapeutic irrigation; subdural space; postoperative complications; mortality
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Trondheim: Burr hole surgery with passive subdural drainage
  Interventions: Procedure: Burr hole surgery with various drainage techniques
- Tromsø: Burr hole surgery with continuous irrigation
  Interventions: Procedure: Burr hole surgery with various drainage techniques
- Stockholm: Burr hole surgery with active subgaleal drainage
  Interventions: Procedure: Burr hole surgery with various drainage techniques

INTERVENTIONS:
Procedure: Burr hole surgery with various drainage techniques — Surgical technique
  1. Continuous irrigation and drainage
  2. Passive subdural drain
  3. Active subgaleal drain

SUMMARY:
There are numerous reported ways to treat chronic subdural hematomas (CSDH) and practice is still differing considerably between departments. Except for a recent randomized controlled trial (RCT) that found that postoperative subdural drainage was better than no drain, there is no higher level evidence. Another recent RCT did not replicate these findings, but the study was severely underpowered.

Aim of this population based study is to compare clinical results (reoperation rates, complications, perioperative death, and survival) between neurosurgical departments treating CSDH with different treatment policies.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with evacuation of primary chronic subdural hematoma(CSDH) from 2005 through 2010 at St.Olav University Hospital
* All patients treated with evacuation of primary chronic subdural hematoma(CSDH) from 2005 through 2010 at University Hospital North Norway
* All patients treated with evacuation of primary CSDH from 2006 through 2010 at Karolinska University Hospital (not 2005 due to practical reasons since major changes occurred in electronic surgery protocols 2005).

Exclusion Criteria:

* Chronic subdural hematoma in arachnoid cyst(s)
* Previous CSDH surgery
* External hydrocephalus (hydrocephalus with cerebrospinal fluid (CSF) in the subdural space rather than in the ventricles)
* CSDH due to previous intracranial surgery (within 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients have been selected to the given therapy solely on the basis of geography. All patients treated with evacuation of primary chronic subdural hematoma(CSDH) from 2005 through 2010 at St.Olav University Hospital and UNN, and primary CSDH from 2006 through 2010 at Karolinska University Hospital (not 2005 due to practical reasons since major changes occurred in electronic surgery protocols 2005).
Sampling Method: Non-Probability Sample
Enrollment: 1258 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
reoperations | 1 year
  Number of reoperations (X/N, %) between centers

SECONDARY OUTCOMES:
continuous irrigation versus other drainage | 1 year
  Number of reoperations with use of continuous irrigation (UNN) versus other drainage (St.Olav, Karolinska)
perioperative death | 30 days
survival | 3 years
  Minimum 3 years follow up. Report 1 year mortality and use of Kaplan Meier curves (log rank test)
surgical complications | 30 days
  As defined by the Ibanez classification where it is the treatment given for a complication that gives the score. Medical and surgical complication is both mentioned and reported seperately

CONTACTS AND LOCATIONS:
Overall Officials: Lars Jacob Stovner, MD PhD, Study Chair — St. Olavs Hospital
Locations (3):
- Norway (2):
  - University Hospital of North Norway, Tromsø
  - St Olavs Hospital, Trondheim
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Result] Sjavik K, Bartek J, Sagberg LM, Henriksen ML, Gulati S, Stahl FL, Kristiansson H, Solheim O, Forander P, Jakola AS. Assessment of drainage techniques for evacuation of chronic subdural hematoma: a consecutive population-based comparative cohort study. J Neurosurg. 2017 Jun 23;133(4):1113-1119. doi: 10.3171/2016.12.JNS161713. PMID 28644099